CLINICAL TRIAL: NCT04390451
Title: Initial Testing of Whole Health STEPS (Structured Tiered Engagement With Peer Support)
Brief Title: Initial Testing of Whole Health STEPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: D3390-W
Record Dates: First submitted 2020-05-13; First posted 2020-05-15 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Mental Health
Keywords: Primary Health Care; Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study compares Whole Health STEPS to a waitlist control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whole Health STEPS (Experimental): Participants will immediately receive Whole Health STEPS.
  Interventions: Behavioral: Whole Health STEPS
- Waitlist (Other): Participants will receive Whole Health STEPS after a defined waiting period.
  Interventions: Behavioral: Whole Health STEPS

INTERVENTIONS:
Behavioral: Whole Health STEPS — A peer-delivered package of Whole Health services.
  Other Names: Whole Health Structured Tiered Engagement with Peer Support

SUMMARY:
This clinical trial is evaluating Whole Health STEPS (Structured Tiered Engagement with Peer Support), a package of services designed to improve functional outcomes for primary care Veterans with mental health concerns who are not actively engaged in mental health services. Whole Health STEPS uses a Peer Support Specialist, or Peer, to provide support for Veterans to make progress on wellness goals using the Whole Health model. The level of support provided will be determined based on Veterans' progress and will be stepped-up until Veterans receive the level of support they need. Whole Health STEPS offers a non-mental health referral option for primary care Veterans with mental health concerns, provides a structured package of existing Whole Health services, and provides a structured service for peers in primary care settings.

ELIGIBILITY:
Inclusion Criteria:

* Veteran status
* Enrolled in primary care at a participating site
* Have at least mild functional impairment
* Screen positive on at least one primary care mental health screener

Exclusion Criteria:

* Actively engaged with an equivalent or higher level of care
* Preference for direct referral to mental health care
* Recent changes to psychotropic medications
* Severe impairment preventing engagement in the intervention or warranting a direct referral to a licensed independent provider
* Inability to independently communicate in verbal and written English
* Inability to complete the research tasks or intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Inventory of Psychosocial Functioning (IPF) | 4 months
  This 80 item self-report inventory measures several domains of psychosocial functioning (e.g., family relationships, work, self-care) on a 0-100 scale with lower scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Emily M. Johnson, PhD, Principal Investigator — Syracuse VA Medical Center, Syracuse, NY
Locations (1):
- Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared upon written request for appropriate scientific reasons.
Supporting Information: SAP
Time Frame: The dataset will be available following publication of the primary manuscript for this project.
Access Criteria: The dataset will be released upon written request for scientific purposes including re-analysis and validation of results.

DOCUMENTS (1):
  • Informed Consent Form (2023-10-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT04390451/ICF_000.pdf